CLINICAL TRIAL: NCT06641973
Title: Technological Balance and Gait Rehabilitation in Patients With Feed and Eating Disorders: Effects on Functional, Motor, and Cognitive Outcomes
Brief Title: Technological Balance Rehabilitation in Feed and Eating Disorders
Acronym: ROAR-FED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6656
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-04

CONDITIONS: Feeding Disorders; Anorexia Nervosa; Bulimia Nervosa
Keywords: Rehabilitation; Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (G-Hun) (Experimental): The experimental group (G-Hun), will carry out robotic balance treatment with the hunova® robotic platform lasting 30 minutes per session, 2 times a week for 5 weeks, in addition to their clinical pathway services.
  Interventions: Device: Robotic balance rehabilitation with hunova® robotic platform
- Control Group (G-Con) (No Intervention)

INTERVENTIONS:
Device: Robotic balance rehabilitation with hunova® robotic platform — The G-Hun will perform robotic balance treatment with the hunova® robotic platform lasting 30 minutes per session, 2 times a week for 5 weeks, in addition to the services provided in their clinical pathway.
  Arms: Experimental Group (G-Hun)

SUMMARY:
Postural control depends on the central integration of vestibular, visual, and somatosensory inputs and the integrity of the neural efferent motor pathway, which continuously provides postural adjustments to environmental and body position changes. It is considered a complex skill and involves the integration of movement strategies necessary for maintaining balance. Decreased postural control can induce instabilities that affect the performance of daily activities and increase the risk of falls. Decreased postural control can be linked to fluctuations in body weight: significant weight gain or loss, in fact, can induce musculoskeletal adaptations , which contribute to postural and motor alterations . In Italy, approximately 3 million people are affected by Feed and Eating Disorders (FED), which include, among others, anorexia nervosa (AN), bulimia nervosa (BN) and uncontrolled eating disorder (UED). There are works in the literature highlighting that both anorexic and obese patients present with impaired postural control and, consequently, reduced balance.

DETAILED DESCRIPTION:
Some authors have pointed out that altered sensitivity may be related to impaired balance and/or postural control in obese patients : in fact, less accurate proprioceptive information is more detrimental to postural stability, especially in more demanding tasks . To prevent balance problems due to impaired proprioception, some authors suggest sensory training . However, to date, there are no works investigating the role of proprioceptive rehabilitation in patients with FED.

The purpose of this study is to evaluate the effects of technological rehabilitation using a robotic platform (hunova® Movendo Technology srl, Genoa, IT) on motor performance, cognitive performance, mood, fatigue, and quality of life.

Patients meeting the inclusion criteria will be recruited from the UOC Clinical and Emergency Psychiatry and the Outpatient Clinics of the Clinical Psychiatry and Addiction Area, and will be evaluated and treated at the UOS Post-Acute Rehabilitation, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy. Patients will be divided into 2 groups by randomization, as specified below. One group (G-Hun), will perform the robotic balance treatment with the robotic platform (hunova®) lasting 30 minutes per session, 2 times a week for 5 weeks, in addition to the services provided by their clinical pathway; while the other group (G-Con), will perform the services provided by the clinical pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Diagnosis of AN, BN, DAI according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders-5 Edition, DSM-5)
* Ability to walk independently or with little assistance;
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Current or past cognitive disorders (mental retardation) with Mini Mental State Evaluation (MMSE) values ≤ 26 ;
* Severe clinical conditions (head trauma, severe neurological and cardiac diseases and vascular disorders, oncological diseases);
* Substance use disorders;
* Unstabilized major psychiatric disorders (e.g., manic episode, acute psychotic episode, etc.);
* Taking medications that alter cardiac activity;
* Orthopedic or postural problems;
* Presence of plantar ulcers;
* Partial or total amputation of foot segments;
* Inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proprioception | Change from Baseline proprioception at 5 weeks
  Improved proprioception as assessed by reduction of Center of Pressure (COP) oscillations using the hunova robotic platform

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Change from Baseline BBS at 5 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Timed Up and Go Test (TUG) | Change from Baseline TUG at 5 weeks
  The Timed Up and Go test (TUG) measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severely abnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from initial getting up to re-seating. Patients are compared with the mean time of adults in their age group, 60 to 69, 70 to 79, and 80 to 99 years of age.
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 5 weeks
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). Three domains, which include balance, usual or self-selected gait speed, and lower limb strength, are assessed by a three-stage balance test (feet side-by-side, semitandem, and tandem positions), a 3-m or 4-m gait speed test (time spent to walk the course), and a repetitive chair stand test (five times chair sit-to-stand test), respectively. A 0- to 12-point scale is used to score the sum of the three assessments with higher point values corresponding with greater levels of physical function and lower disability, whereas lower point values correspond with lower levels of physical function and higher disability, respectively.
Timed-25 Foot Walk (T25FW) | Change from Baseline T25FW at 5 weeks
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Mental Deterioration battery (MDB) | Change from Baseline MDB at 5 weeks
  The MDB is a neuropsychological test battery for detecting mental deterioration and comprises 7 tests divided into verbal and visuospatial tests, which can be administered independently of each other.
  VERBAL TESTS are: immediate and delayed recall of Rey's 15 words, phonological verbal fluency; sentence construction VISUAL-SPACE TESTS are: Raven's coloured progressive matrices (PM47; immediate visual memory; copying of freehand drawings) All MDB tests are corrected using the Equivalent Scores method, after correction for factors (age, years of schooling) of the score obtained.
Trial Making Test (TMT) | Change from Baseline TMT at 5 weeks
  The Trail Making Test (TMT) measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of Thumb Most in 90 seconds Trail B: Average 75 seconds, Deficient > 273 seconds, Rule of Thumb Most in 3 minutes
Symbol Digit Modalities Test (SDMT) | Change from Baseline SDMT at 5 weeks
  The Symbol Digit Modalities Test (SDMT) is a test that assesses information processing speed and consists of a series of nine printed symbols to which nine numbers correspond. After a 'training' phase, patients are asked to match as many symbols as possible to the corresponding number in just 90 seconds. As the test persons can give written or oral answers, the test is suitable for people with motor disabilities or speech disorders.
  The score is calculated by adding up the number of correct substitutions in the 90-second interval (maximum = 110). Interpretation results from normalising the categories of gender, age and education.
Stroop Colour Word Test (SCWT) | Change from Baseline SCWT at 5 weeks
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task, to name colors in the second and third tasks. It is necessary to mark both any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Eating Disorder Inventory (EDI-3) | Change from Baseline EDI-3 at 5 weeks
  The EDI-3 is an instrument for self-assessment of symptoms commonly associated with anorexia and bulimia. It contains 91 items divided into twelve subscales assessed by a 0-4 point scoring system. Three EDI-3 items are specific to eating disorders, while 9 are general psychological scales relevant to eating disorders. The inventory produces six composite scores: eating disorder risk, ineffectiveness, interpersonal problems, affective problems, hypercontrol, and general psychological maladjustment.
  Higher values indicate a worse condition
Eating Disorder Examination Questionnaire 7.0 (EDE-Q) | Change from Baseline EDE-Q at 5 weeks
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire that assesses the range, frequency, and severity of behaviors associated with an eating disorder diagnosis. It is divided into 4 subscales (Restriction, Eating Concern, Fitness Concern, and Weight Concern) and an overall score; a higher score indicates more problematic eating difficulties.
  Higher values indicate a worse condition.
Binge-Eating Scale (BES) | Change from Baseline BES at 5 weeks
  The Binge Eating Scale (BES) is a self-report instrument developed to assess the presence and behavioral manifestations of Binge Eating Disorder (BED). Consisting of 16 items, the BES assesses both the severity and frequency of binge eating episodes, which are critical to diagnosing and understanding the disorder.
  Higher values indicate a worse condition.
Heartbeat Perception Task (HPT) | Change from Baseline HPT at 5 weeks
  HPT is a method used to assess an individual's interoceptive accuracy or ability to perceive internal bodily sensations accurately. Higher values indicate a worse condition.
Depression Anxiety Stress Scales Short Version (DASS-21) | Change from Baseline DASS-21 at 5 weeks
  DASS-21 is a depression, anxiety and stress assessment scale consisting of 21 items. Participants are asked to indicate how much the statement applies to them in reference to the previous week on a 4-point Likert scale (from 0 = Does not apply at all to me to 3 = Applies a lot or most of the time to me). It allows for the detection of three dimensions: Depression (item example: "I felt like I had nothing to look forward to"), Anxiety (item example: "I felt close to a panic attack"), Stress (item example: "I found it hard to relax"). Higher values indicate a worse condition.
Difficulties in Emotion Regulation Scale-2 (DERS) | Change from Baseline DERS at 5 weeks
  DERS is an instrument that measures emotion regulation problems. The 36-item self-report scale asks respondents how they relate to their emotions to produce scores on the following subscales.
  (i) Non-acceptance of emotional responses (ii) Difficulty engaging in goal-oriented behaviors (iii) Difficulty controlling impulses (iv) Lack of emotional awareness (v) Limited access to emotion regulation strategies (vi) Lack of emotional clarity Scores are presented as total scores and as scores for each of the 6 subscales. Higher scores indicate greater problems with emotion regulation.
Body Uneasiness Test (BUT) | Change from Baseline BUT at 5 weeks
  The BUT is a 71-item self-report questionnaire divided into two parts: BUT-A, which measures weight phobia, concerns about body image, avoidance, compulsive self-monitoring, and feelings of detachment and estrangement toward one's body (depersonalization); and BUT-B, which examines specific concerns about particular body parts or functions.
  The BUT consists of 34 items on a Lickert scale of 0 to 5 classifiable into 5 scales (weight phobia, body image preoccupation, compulsive self-monitoring, avoidance, and depersonalization). Higher values indicate a worse condition.
Toronto Alexithymia Scale 20-item version (TAS-20) | Change from Baseline TAS-20 at 5 weeks
  The TAS-20 is a 20-item self-administered questionnaire that measures the difficulty in identifying and describing emotions, which is an important part of alexithymia. For each item there is a choice of 5 responses: Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree. Each item is rated on a 5-point Likert-type scale (1 = strongly disagree; 5 = strongly agree). Scoring range: 20-100 (higher scores indicate greater difficulty). The TAS-20 uses a cutoff score: 0-51=No alexithymia, 52-60=Possible alexithymia, and 61-100=Alexithymia present.
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 5 weeks
  The Modified Fatigue Impact Scale (MFIS) is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
EuroQoL- 5D (EQ-5D) | Change from Baseline EQ-5D at 5 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Silver Index (SI) | Change from Baseline SI at 5 weeks
  The SI is an objective test to identify the risk of falling, which is carried out using the Hunova robotic platform. It consists of seven domains:
  (i) static balance (ii) dynamic balance (iii) reactive balance (iv) sensory integration (v) stability limits (vi) sitting-to-standing position (vii) gait speed. At the end of the evaluation you get a percentage that indicates the risk of falling

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No